CLINICAL TRIAL: NCT01618669
Title: A Phase 3b, Open-Label, Parallel Group, Randomized, Multicenter Study to Assess Regadenoson Administration Following an Inadequate Exercise Stress Test as Compared to Regadenoson Alone for Myocardial Perfusion Imaging (MPI) Using Single Photon Emission Computed Tomography (SPECT)
Brief Title: A Study to Assess Regadenoson Administration Following an Inadequate Exercise Stress Test as Compared to Regadenoson Alone for Myocardial Perfusion Imaging (MPI) Using Single Photon Emission Computed Tomography (SPECT)
Acronym: EXERRT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 3606-CL-3004
Record Dates: First submitted 2012-05-29; First posted 2012-06-13 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: Coronary Artery Disease (CAD); regadenoson; pharmacologic stress
MeSH Terms: conditions — Coronary Artery Disease | interventions — regadenoson

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regadenoson After Peak Exercise (Experimental): On Day 1 participants received regadenoson, 0.4 mg in a 5 mL intravenous bolus, 3 minutes after exercise while in walk recovery and then a stress SPECT MPI. One to 14 days later participants received regadenoson at rest and then a stress SPECT MPI.
  Interventions: Drug: Regadenoson; Procedure: Single photon emission computed tomography (SPECT) myocardial perfusion imaging (MPI)
- Regadenoson Alone (Active Comparator): On Day 1 participants received regadenoson, 0.4 mg in a 5 mL intravenous bolus (1 hour after exercise recovery), and then stress SPECT MPI. One to 14 days later participants received regadenoson at rest and then a stress SPECT MPI.
  Interventions: Drug: Regadenoson; Procedure: Single photon emission computed tomography (SPECT) myocardial perfusion imaging (MPI)

INTERVENTIONS:
Drug: Regadenoson — Administered as an intravenous (IV) bolus
  Other Names: Lexiscan; CVT3146
Procedure: Single photon emission computed tomography (SPECT) myocardial perfusion imaging (MPI)

SUMMARY:
The purpose of this study is to demonstrate that the strength of agreement between single photon emission computed tomography (SPECT) imaging with regadenoson following inadequate exercise stress testing and SPECT imaging with regadenoson alone is not inferior to the strength of agreement between two sequential regadenoson SPECT images without exercise.

ELIGIBILITY:
Inclusion Criteria:

* Subjects referred for an exercise or pharmacologic stress test SPECT MPI procedure for the evaluation of coronary artery disease (CAD) are eligible for study participation. Subjects referred for pharmacologic stress should have a reasonable potential of attempting exercise stress. Subject must have one of the following:

  * a. Past ischemia on any prior imaging stress test without invasive intervention on the artery subtending this territory
  * b. Subject with known CAD who have symptoms similar to previous ischemic symptoms, or recent onset of symptoms or recently worsened symptoms suggestive of ischemia
  * c. Diamond Forrester estimated pretest probability of CAD of ≥ 50%
  * d. History of most recent coronary artery bypass surgery or most recent percutaneous coronary intervention (PCI) > 10 years (patients who are > 30 days but less than 10 years post coronary artery bypass graft (CABG) or PCI can be included if they meet criteria a, b, or e)
  * e. Previously demonstrated 100% occlusion by invasive coronary or computed tomography (CT) angiography without successful intervening revascularization as these foods may alter regadenoson effects

Exclusion Criteria:

* Subject has a clinically significant illness, medical condition, or laboratory abnormality
* Female subject who is pregnant or lactating
* Subject is on dialysis for end stage renal disease or has a history of glomerular filtration rate (GFR) < 15 mL/min (calculated using MDRD [Modification of Diet in Renal Disease] formula)
* Subject has a history of coronary revascularization by either PCI or CABG within 1 month prior to the rest myocardial perfusion imaging (MPI)
* Subject has a pacemaker or an implantable cardioverter defibrillator (ICD)
* Subject has a history of acute myocardial infarction (MI) or high risk unstable angina within 30 days prior to the rest MPI or has had cardiac transplantation
* Subject has uncontrolled hypertension at any point on Visit 2 prior to exercise testing (i.e., systolic blood pressure (SBP) ≥ 180 or diastolic blood pressure (DBP) ≥ 95 mmHg on two consecutive measurements while at rest).
* Subject has severe aortic stenosis or hypertrophic cardiomyopathy with obstruction or has decompensated congestive heart failure
* Subject has a history of severe respiratory disease including: asthma, chronic obstructive pulmonary disease (COPD) or other bronchospastic reactive airway disease or who is on 24-hour continuous oxygen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1147 (Actual)
Dates: Start 2012-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (69):
- United States (60):
  - Mobile Heart Specialists, PC, Mobile, Alabama
  - Silicon Valley Medical Imaging, Fremont, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - Westside Medical Associates of Los Angeles, Los Angeles, California
  - Ventura Clinical Trials, Malibu, California
  - Mission Internal Medical Group, Mission Viejo, California
  - VA San Diego Healthcare System, San Diego, California
  - Santa Rosa Cardiology Medical Group, Inc., Santa Rosa, California
  - Los Angeles Biomedical Research Institute, Torrance, California
  - HOCC - New Britain Campus, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfieri Cardiology, Newark, Delaware
  - Delaware Clinical Trials, Wilmington, Delaware
  - Elite Research and Clinical Trials, Aventura, Florida
  - S & W Clinical Research, Fort Lauderdale, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Florida Heart Associates, Fort Myers, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - St. Luke's Cardiology St. Vincent's HealthCare, Jacksonville, Florida
  - Watson Medical Clinic/Lakeland Regional Medical Clinic, Lakeland, Florida
  - MIMA Century Research Associates, Melbourne, Florida
  - Cardiovascular Research Center of South Florida, Miami, Florida
  - Florida Hospital/Cardiovascular Institute, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - St. Joseph's Hospital, Atlanta, Georgia
  - University Cardiology Associates, LLC, Augusta, Georgia
  - South Coast Medical Group, Savannah, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - I U School of Medicine/ Krannert Institute of Cardiology, Indianapolis, Indiana
  - Midwest Cardiology Associates, Overland Park, Kansas
  - Maine Research Associates, Portland, Maine
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Berkshire Medical Center, Pittsfield, Massachusetts
  - Henry Ford Hospital, Detriot, Michigan
  - Wayne State University, Detroit, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Cardiology Associates of North Mississippi, Tupelo, Mississippi
  - Cardiovascular Imaging Technologies, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Alegent Health Heart and Vascular Specialists, Omaha, Nebraska
  - Alegent Health Research Center, Omaha, Nebraska
  - Las Vegas Radiology, Las Vegas, Nevada
  - Laurelton Medical center, Laurelton, New York
  - Columbia University Medical Center, New York, New York
  - Westchester Medical Center-New York Medical College, Valhalla, New York
  - Buffalo Cardiology & Pulmonary Associates, P.C., Williamsville, New York
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Berks Cardiologists, Ltd., Wyomissing, Pennsylvania
  - Katy Cardiology Associates, Katy, Texas
  - Mission Research Institute LLC, New Braunfels, Texas
  - West Houston Area Clinical Trial Consultants, LLC, Tomball, Texas
  - University of Virginia, Charlottesville, Virginia
  - Roanoke Heart Institute, PC, Roanoke, Virginia
  - University of Washington, Seattle, Washington
- Argentina (5):
  - Hospital Italiano Garibaldi, Rosario, Santa Fe Province
  - Instituto Oulton, Córdoba
  - Instituto de Cardiologia la Plata, La Plata
  - Hospital Italiano de La Plata, Provincia de Buenos Aires
  - Sanatorio San Geronimo, Santa Fe
- Peru (3):
  - Clinica Anglo Americana, Lima
  - Hospital Arzobispo Loayza, Lima
  - Instituto Nacional Cardiovascular de EsSalud, Lima
- VA Caribbean Healthcare System (672), San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Thomas GS, Cullom SJ, Kitt TM, Feaheny KM, Ananthasubramaniam K, Gropler RJ, Jain D, Thompson RC. The EXERRT trial: "EXErcise to Regadenoson in Recovery Trial": A phase 3b, open-label, parallel group, randomized, multicenter study to assess regadenoson administration following an inadequate exercise stress test as compared to regadenoson without exercise for myocardial perfusion imaging using a SPECT protocol. J Nucl Cardiol. 2017 Jun;24(3):788-802. doi: 10.1007/s12350-017-0813-3. Epub 2017 Feb 21. PMID 28224449
- See also: Link to results on Astellas Clinical Study Results Web site — https://www.astellasclinicalstudyresults.com/study.aspx?ID=3606-CL-3004

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 49 sites in a total of 3 countries including the United States (44 sites), Argentina (4 sites) and Peru (1 site).
Pre-assignment Details: At Baseline, patients meeting all inclusion/exclusion criteria completed single photon emission computed tomography (SPECT) myocardial perfusion imaging (MPI) while at rest. Participants then underwent a Bruce or modified Bruce exercise protocol; those unable to reach 85% maximum predicted heart rate and/or 5 metabolic equivalents were randomized.
Groups:
- Regadenoson After Peak Exercise: On Day 1 participants received regadenoson, 0.4 mg in a 5 mL intravenous bolus, 3 minutes after exercise while in walk recovery and then a stress SPECT myocardial perfusion imaging (MPI). One to 14 days later participants received regadenoson at rest and then a stress SPECT MPI.
- Regadenoson Alone: On Day 1 participants received regadenoson, 0.4 mg in a 5 mL intravenous bolus, (1 hour after exercise recovery) and then stress SPECT MPI. One to 14 days later participants received regadenoson at rest and then a stress SPECT MPI.
Period: Overall Study
Arm/Group | Regadenoson After Peak Exercise | Regadenoson Alone
Started | 578 | 569
Received Treatment | 575 | 567
Completed | 544 | 546
Not Completed | 34 | 23
Not completed — Lost to Follow-up | 1 | 1
Not completed — Randomized but Never Received Study Drug | 3 | 2
Not completed — Adverse Event | 16 | 7
Not completed — Protocol Violation | 5 | 3
Not completed — Withdrawal by Subject | 9 | 9
Not completed — Miscellaneous Reason | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who took at least 1 dose of study drug (Safety Analysis Set).
Groups:
- Total: Total of all reporting groups
Arm/Group | Regadenoson After Peak Exercise | Regadenoson Alone | Total
Number analyzed (Participants) | 575 | 567 | 1142
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (11.45) | 61.9 (11.19) | 61.9 (11.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 234 | 239 | 473
  Male | 341 | 328 | 669
Bruce Exercise Group [Number; unit: participants] — The Bruce exercise test involves walking on a treadmill while the heart is monitored by an electrocardiograph. The protocol consists of several stages of progressively greater workloads.
  The Modified Bruce protocol starts at a lower workload than the standard test and is typically used for elderly or sedentary patients.
  Data are reported for all randomized participants with interpretable SPECT scans at all visits as determined by at least 2 of the 3 blinded independent expert readers (full analysis set; 538 and 534 participants in each treatment group respectively).
  participants
    Standard Bruce Exercise | 448 | 442 | 890
    Modified Bruce Exercise | 90 | 93 | 183
Maximum Metabolic Equivalents Achieved [Mean (Standard Deviation); unit: metabolic equivalents] — A metabolic unit used to quantify the intensity of physical activity, which is defined as the ratio of the metabolic rate during exercise to the metabolic rate at rest. One MET corresponds to an energy expenditure of approximately 1 kcal/kg/hour, or an oxygen uptake of 3.5 ml of O2 consumption/kg/hour.
  Data are provided for the full analysis set (538 and 534 participants in each treatment group respectively).
  metabolic equivalents | 5.45 (2.284) | 5.37 (2.331) | 5.41 (2.307)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Majority Reader Self-agreement in Ischemia Assessment Between First and Second Stress Scans
Description: SPECT scans were reviewed in a blinded fashion by 3 independent expert readers using the 17-segment model for standardized myocardial segmentation. At rest and stress, each segment was scored on a 0 (normal) to 4 (absent contrast/radiotracer uptake) scale by each of the 3 blinded readers according to the amount of contrast or radiotracer the myocardium in the segment absorbed. If the stress score was ≥ 2 and the rest score was less than the stress score, the segment was counted as having a reversible defect.
  The number of segments with reversible defects was categorized as absence (0 - 1 reversible segments) or presence (≥ 2 defects reversible segments) of ischemia.
  Each reader was defined as having self-agreement based upon identical categorization of a given participant as absent or present for ischemia for both the initial and second stress visits.
  Majority agreement is if at least 2 out of the 3 blinded readers demonstrated self-agreement for a given participant.
Time Frame: Day 1 (rest scan and first stress scan) and Day 2 -15 (second stress scan)
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Regadenoson After Peak Exercise | Regadenoson Alone
Number analyzed (Participants) | 538 | 535
proportion of participants | 0.92 [0.89 to 0.94] | 0.95 [0.93 to 0.97]
Statistical Analysis 1: Comparison: Regadenoson After Peak Exercise vs Regadenoson Alone; Test type: Non-Inferiority or Equivalence — If the lower confidence bound of the 1-sided alpha level of 0.025 of the difference in the proportion of participants with majority reader self-agreement exceeded -0.075, non-inferiority would be demonstrated; Difference = -0.03, 95% CI 2-sided [-0.06 to -0.00], Standard Error of Mean 0.015 — Difference equals Regadenoson After Peak Exercise minus Regadenoson Alone

2. Secondary Outcome: Percentage of Participants With Treatment-emergent Clinically Significant Cardiac Events
Description: A clinically significant cardiac event is defined as:
  * Any of the following events found on the Holter electrocardiogram (ECG)/12-Lead ECG within 1 hour after regadenoson administration:
    * ventricular arrhythmias (sustained ventricular tachycardia, ventricular fibrillation, torsade de pointes, ventricular flutter),
    * ST-T depression (> 2 mm),
    * ST-T elevation (≥1 mm),
    * Atrioventricular (AV) block (2:1 AV block, AV Mobitz I, AV Mobitz II, complete heart block)
    * sinus arrest > 3 seconds in duration
  Or
  * a treatment-emergent adverse event (TEAE) per the Medical Dictionary for Regulatory Activities (MedDRA) Standardised MedDRA Queries (SMQ) (Narrow Scope) for myocardial infarction
  Or
  * a TEAE preferred term of angina unstable within 24 hours of regadenoson administration.
Time Frame: Within 1 hour for ECG events and up to 24 hours for adverse events after administration of regadenoson
Population: Safety analysis set (all randomized participants who received at least 1 dose of regadenoson study drug)
Measure: Number; unit: percentage of participants
Groups:
- Regadenoson After Peak Exercise: MPI 1; Regadenoson After Peak Exercise: MPI 2: On Day 1 participants received regadenoson, 0.4 mg in a 5 mL intravenous bolus, 3 minutes after exercise while in walk recovery and then a stress SPECT MPI. One to 14 days later participants received regadenoson at rest and then a stress SPECT MPI.
- Regadenoson Alone: MPI 1; Regadenoson Alone: MPI 2: On Day 1 participants received regadenoson, 0.4 mg in a 5 mL intravenous bolus, (1 hour after exercise recovery) and then stress SPECT MPI. One to 14 days later participants received regadenoson at rest and then a stress SPECT MPI.
Arm/Group | Regadenoson After Peak Exercise: MPI 1 | Regadenoson After Peak Exercise: MPI 2 | Regadenoson Alone: MPI 1 | Regadenoson Alone: MPI 2
Number analyzed (Participants) | 575 | 544 | 567 | 548
percentage of participants
  Any Event | 3.0 | 0.9 | 0.5 | 0.4
  Any Holter/12-Lead ECG Abnormality | 2.8 | 0.9 | 0.5 | 0.4
  Sustained Ventricular Tachycardia | 0.0 | 0.0 | 0.0 | 0.0
  Ventricular Fibrillation or Ventricular Flutter | 0.0 | 0.0 | 0.0 | 0.0
  Torsade de Pointes | 0.0 | 0.0 | 0.0 | 0.0
  ST-T Depression (≥ 2 mm) | 2.3 | 0.6 | 0.4 | 0.4
  ST-T Elevation (≥ 1 mm) | 0.5 | 0.4 | 0.2 | 0.0
  2:1 AV Block | 0.0 | 0.0 | 0.0 | 0.0
  Mobitz I Second Degree AV Block | 0.0 | 0.0 | 0.0 | 0.0
  Mobitz II Second Degree AV Block | 0.0 | 0.0 | 0.0 | 0.0
  Complete Heart Block | 0.0 | 0.0 | 0.0 | 0.0
  Pause > 3.0 seconds | 0.0 | 0.0 | 0.0 | 0.0
  Any TEAE per SMQ for Myocardial Infarction | 0.3 | 0.0 | 0.0 | 0.0
  Acute Coronary Syndrome | 0.2 | 0.0 | 0.0 | 0.0
  Myocardial Infarction | 0.2 | 0.0 | 0.0 | 0.0
  Adverse Event of Angina Unstable | 0.0 | 0.0 | 0.0 | 0.0

3. Secondary Outcome: Proportion of Participants With Agreement in the Assessment of Absence or Presence of Ischemia Between First and Second Stress Scans
Description: The number of segments with reversible defects was assessed by each of the 3 blinded independent expert readers. Based on the median count of the number of reversible defects across the 3 readers, categorized as absence (0 to 1 reversible segments) or presence (≥ 2 reversible defects) of ischemia, the proportion of participants with agreement in the presence and absence of ischemia between the first and second stress scans was calculated.
Time Frame: Day 1 (stress MPI 1) and Day 2 -15 (stress MPI 2)
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Regadenoson After Peak Exercise | Regadenoson Alone
Number analyzed (Participants) | 538 | 535
proportion of participants | 0.75 [0.68 to 0.83] | 0.77 [0.67 to 0.86]
Statistical Analysis 1: Comparison: Regadenoson After Peak Exercise vs Regadenoson Alone; Test type: Non-Inferiority or Equivalence — The lower confidence bound of the 1-sided alpha level of 0.025 of the difference in agreement rates must exceed -0.10 in order to demonstrate non-inferiority; Difference = -0.01, 95% CI 2-sided [-0.14 to 0.11], Standard Error of Mean 0.063 — Difference equals Regadenoson After Peak Exercise minus Regadenoson Alone

4. Secondary Outcome: Proportion of Participants With Agreement in the Assessment of Reversible Defects in 3 Categories of Ischemia Between First and Second Stress Scans
Description: The number of segments with reversible defects was assessed by each of the 3 blinded independent expert readers. Based on the median count of the number of reversible defects across the 3 readers, categorized as 0 to 1, 2 to 4, or ≥ 5 reversible segments, the proportion of participants with agreement in the three ischemia categories between the first and second stress scans was to be calculated. In the reported data, these proportions only include the 0-1 and 2-4 categories; the ≥ 5 category was not included because there were no participants in this category for the Regadenoson Alone group for the initial stress MPI.
Time Frame: Day 1 (stress MPI 1) and Day 2 - 15 (stress MPI 2)
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Regadenoson After Peak Exercise | Regadenoson Alone
Number analyzed (Participants) | 538 | 535
proportion of participants | 0.73 [0.69 to 0.77] | 0.75 [0.71 to 0.78]
Statistical Analysis 1: Comparison: Regadenoson After Peak Exercise vs Regadenoson Alone; Test type: Non-Inferiority or Equivalence — The lower confidence bound of the 1-sided alpha level of 0.025 of the difference in agreement rates must exceed -0.133 in order to demonstrate non-inferiority. Non-inferiority could not be assessed because of insufficient data in the Regadenoson Alone group; Difference = -0.02, 95% CI 2-sided [-0.07 to 0.04], Standard Error of Mean 0.027

5. Secondary Outcome: Proportion of Participants With Agreement in the Summed Stress Score (SSS) Between First and Second Stress Scans
Description: The 17-segment model for standardized myocardial segmentation was used to analyze MPI scans. Each segment was scored on a 0 to 4 scale according to the amount of contrast or radiotracer the myocardium in the segment absorbed:
  * 0: normal perfusion
  * 1: slightly reduced contrast/radiotracer uptake
  * 2: moderately reduced contrast/radiotracer uptake
  * 3: severely reduced contrast/radiotracer uptake
  * 4: absent contrast/radiotracer uptake.
  The Summed Stress Score (SSS) was calculated as the sum of the stress scores across the 17 segments. The mean value (rounded to the nearest integer) across the 3 readers was computed and the SSS was categorized into 4 group categorical variables based on the score: 0 to 3, 4 to 7, 8 to 11, and ≥ 12. The proportion of participants with agreement in respect to these categories between the two stress scans was calculated.
Time Frame: Day 1 (stress MPI 1) and Day 2 - 15 (stress MPI 2)
Population: Full Analysis Set
Measure: Number; unit: proportion of participants
Arm/Group | Regadenoson After Peak Exercise | Regadenoson Alone
Number analyzed (Participants) | 538 | 535
proportion of participants | 0.86 | 0.84
Statistical Analysis 1: Comparison: Regadenoson After Peak Exercise vs Regadenoson Alone; Test type: Superiority or Other; Difference = 0.02, 95% CI 2-sided [-0.03 to 0.06], Standard Error of Mean 0.022

6. Secondary Outcome: Proportion of Participants With Agreement in the Summed Difference Score (SDS) Between First and Second Stress Scans
Description: The 17-segment model for standardized myocardial segmentation was used to analyze MPI scans. At rest and stress, each segment was scored on a 0 to 4 scale according to the amount of contrast or radiotracer the myocardium in the segment absorbed:
  * 0: normal perfusion
  * 1: slightly reduced contrast/ uptake
  * 2: moderately reduced contrast/uptake
  * 3: severely reduced contrast/uptake
  * 4: absent contrast/uptake.
  SSS was calculated as the sum of the stress scores across the 17 segments and the Summed Rest Score (SRS) was calculated as the sum of the rest scores across the 17 segments. The Summed Difference Score (SDS) is the difference in the SSS and SRS (SSS - SRS).
  The mean value (rounded to the nearest integer) across the 3 readers was computed and the SDS was categorized into 3 categorical variables based on the score: 0 to 6, 7 to 13 and ≥ 14. The proportion of participants with agreement in respect to these categories between the two stress scans was calculated.
Time Frame: Day 1 (rest MPI and stress MPI 1) and Day 2 - 15 (stress MPI 2)
Population: Full Analysis Set
Measure: Number; unit: participants
Groups:
- REG APEX: MPI 2 SDS 0-6: Participants in the Regadenoson After Peak Exercise (APEX) group who had an SDS from 0 to 6 on their second stress scan.
- REG APEX: MPI 2 7-13: Participants in the Regadenoson After Peak Exercise (REG APEX) group who had an SDS from 7 to 13 on their second stress scan.
- REG APEX: MPI 2 SDS ≥ 14: Participants in the Regadenoson After Peak Exercise (REG APEX) group who had an SDS ≥ 14 on their second stress scan.
- REG Alone: MPI 2 SDS 0-6: Participants in the Regadenoson (REG) Alone group who had an SDS from 0 to 6 on their second stress scan.
- REG Alone: MPI 2 SDS 7-13: Participants in the Regadenoson (REG) Alone group who had an SDS from 7 to 13 on their second stress scan.
- REG Alone: MPI 2 SDS ≥ 14: Participants in the Regadenoson (REG) Alone group who had an SDS ≥ 14 on their second stress scan.
Arm/Group | REG APEX: MPI 2 SDS 0-6 | REG APEX: MPI 2 7-13 | REG APEX: MPI 2 SDS ≥ 14 | REG Alone: MPI 2 SDS 0-6 | REG Alone: MPI 2 SDS 7-13 | REG Alone: MPI 2 SDS ≥ 14
Number analyzed (Participants) | 538 | 538 | 538 | 535 | 535 | 535
participants
  MPI 1 SDS 0-6 | 531 | 4 | 0 | 527 | 3 | 0
  MPI 1 SDS 7-13 | 0 | 3 | 0 | 2 | 3 | 0
  MPI 1 SDS ≥ 14 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Participants With Less, the Same, or More Reversible Perfusion Defects Shown by the First Stress Scan When Compared to the Second Stress Scan
Description: Each reader evaluated the initial stress SPECT MPI scan compared to the participant's second stress SPECT MPI scan (blinded at time of the evaluation) for whether there was Less (-1), the Same (0) or More (1) reversible perfusion defects. The median assessment of the 3 blinded readers was used to summarize the number of participants in each category.
Time Frame: Day 1 (stress MPI 1) and Day 2-15 (stress MPI 2)
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Regadenoson After Peak Exercise | Regadenoson Alone
Number analyzed (Participants) | 538 | 535
participants
  Less Reversible Perfusion Defects | 57 | 49
  Same Number of Reversible Perfusion Defects | 441 | 459
  More Reversible Perfusion Defects | 40 | 27

8. Secondary Outcome: Overall Assessment of Image Quality
Description: The image quality for each scan was rated by each independent reader as 1 = Poor, 2 = Fair, 3 = Good, 4 = Excellent. Based on the median rating of overall image quality across the three readers, the number of participants with each rating is reported for each scan.
Time Frame: Day 1 (rest MPI and stress MPI 1) and Day 2 - 15 (stress MPI 2)
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Regadenoson After Peak Exercise | Regadenoson Alone
Number analyzed (Participants) | 538 | 535
participants
  Rest MPI: Excellent | 140 | 157
  Rest MPI: Good | 307 | 308
  Rest MPI: Fair | 91 | 70
  Rest MPI: Poor | 0 | 0
  Stress MPI 1: Excellent | 224 | 211
  Stress MPI 1: Good | 287 | 291
  Stress MPI 1: Fair | 27 | 33
  Stress MPI 1: Poor | 0 | 0
  Stress MPI 2: Excellent | 192 | 205
  Stress MPI 2: Good | 303 | 293
  Stress MPI 2: Fair | 43 | 37
  Stress MPI 2: Poor | 0 | 0

9. Secondary Outcome: Target to Background Radiotracer Uptake Ratios From the First and Second Stress Scans
Description: Image quality was assessed through radiotracer uptake in the heart (target organ) compared to liver, gut and combined liver plus gut (background interference).
Time Frame: Day 1 (stress MPI 1) and Day 2 - 15 (stress MPI 2)
Population: Full analysis set participants who have planar images available for each scan
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Regadenoson After Peak Exercise: MPI 1 | Regadenoson After Peak Exercise: MPI 2 | Regadenoson Alone: MPI 1 | Regadenoson Alone: MPI 2
Number analyzed (Participants) | 514 | 525 | 518 | 523
ratio
  Heart-to-Liver | 1.05 (0.399) | 0.94 (0.373) | 0.96 (0.365) | 0.95 (0.362)
  Heart-to-Gut | 1.12 (0.436) | 0.99 (0.399) | 1.05 (0.428) | 0.99 (0.387)
  Heart-to-(Liver/Gut) | 1.02 (0.296) | 0.90 (0.260) | 0.94 (0.274) | 0.91 (0.259)

10. Secondary Outcome: Percentage of Scans With Subdiaphragmatic Interference
Description: Each reader assessed the sub-diaphragmatic radiotracer interference with cardiac image quality using a 4-point scale of 0 = none, 1 = slight, 2 = moderate or 3 = severe for each stress SPECT MPI. The median rating across the 3 readers was used to summarize the percentage of scans with interference.
Time Frame: Day 1 (stress MPI 1) and Day 2 -15 (stress MPI 2)
Population: Full Analysis Set
Measure: Number; unit: percentage of stress MPI scans
Arm/Group | Regadenoson After Peak Exercise: MPI 1 | Regadenoson After Peak Exercise: MPI 2 | Regadenoson Alone: MPI 1 | Regadenoson Alone: MPI 2
Number analyzed (Participants) | 284 | 284 | 270 | 270
percentage of stress MPI scans
  None | 0.4 | 0.0 | 0.0 | 0.0
  Slight | 71.8 | 63.7 | 68.1 | 67.4
  Moderate | 27.5 | 36.3 | 31.5 | 32.6
  Severe | 0.4 | 0.0 | 0.4 | 0.0

11. Secondary Outcome: Percentage of Cardiac Segments Obscured by Subdiaphragmatic Activity
Description: The number of cardiac segments obscured by the sub-diaphragmatic activity by group by stress SPECT MPI scan and by reader is reported.
Time Frame: Day 1 (stress MPI 1) and Day - 15 (stress MPI 2)
Population: Full Analysis Set
Measure: Number; unit: percentage of segments
Arm/Group | Regadenoson After Peak Exercise: MPI 1 | Regadenoson After Peak Exercise: MPI 2 | Regadenoson Alone: MPI 1 | Regadenoson Alone: MPI 2
Number analyzed (Participants) | 538 | 538 | 535 | 535
percentage of segments
  Reader 1: Segment 1 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 1: Segment 2 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 1: Segment 3 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 1: Segment 4 | 33.6 | 37.2 | 34.2 | 37.4
  Reader 1: Segment 5 | 9.7 | 8.4 | 7.9 | 7.7
  Reader 1: Segment 6 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 1: Segment 7 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 1: Segment 8 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 1: Segment 9 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 1: Segment 10 | 31.6 | 35.5 | 32.3 | 36.3
  Reader 1: Segment 11 | 9.5 | 8.2 | 7.5 | 7.5
  Reader 1: Segment 12 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 1: Segment 13 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 1: Segment 14 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 1: Segment 15 | 1.7 | 0.9 | 2.4 | 2.1
  Reader 1: Segment 16 | 0.0 | 0.0 | 0.2 | 0.2
  Reader 1: Segment 17 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 2: Segment 1 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 2: Segment 2 | 0.0 | 0.0 | 0.2 | 0.0
  Reader 2: Segment 3 | 0.0 | 0.0 | 0.2 | 0.6
  Reader 2: Segment 4 | 34.4 | 35.1 | 32.5 | 32.5
  Reader 2: Segment 5 | 1.1 | 0.4 | 0.7 | 0.7
  Reader 2: Segment 6 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 2: Segment 7 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 2: Segment 8 | 0.0 | 0.2 | 0.0 | 0.0
  Reader 2: Segment 9 | 0.0 | 0.0 | 0.4 | 0.4
  Reader 2: Segment 10 | 12.6 | 11.9 | 13.8 | 13.1
  Reader 2: Segment 11 | 0.0 | 0.2 | 0.6 | 0.2
  Reader 2: Segment 12 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 2: Segment 13 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 2: Segment 14 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 2: Segment 15 | 9.1 | 8.7 | 10.5 | 9.5
  Reader 2: Segment 16 | 0.0 | 0.2 | 0.0 | 0.0
  Reader 2: Segment 17 | 0.4 | 0.0 | 0.0 | 0.0
  Reader 3: Segment 1 | 0.0 | 0.2 | 0.0 | 0.0
  Reader 3: Segment 2 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 3: Segment 3 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 3: Segment 4 | 14.1 | 16.7 | 17.9 | 17.2
  Reader 3: Segment 5 | 0.6 | 0.4 | 0.7 | 0.2
  Reader 3: Segment 6 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 3: Segment 7 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 3: Segment 8 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 3: Segment 9 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 3: Segment 10 | 16.0 | 17.8 | 18.5 | 18.9
  Reader 3: Segment 11 | 0.7 | 0.2 | 0.6 | 0.2
  Reader 3: Segment 12 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 3: Segment 13 | 0.2 | 0.0 | 0.0 | 0.0
  Reader 3: Segment 14 | 0.0 | 0.0 | 0.0 | 0.0
  Reader 3: Segment 15 | 13.9 | 13.8 | 13.1 | 14.6
  Reader 3: Segment 16 | 0.4 | 0.7 | 0.4 | 0.2
  Reader 3: Segment 17 | 0.9 | 0.9 | 0.7 | 0.6

12. Secondary Outcome: Number of Participants With Adverse Events Within 24 Hours After Administration of Regadenoson
Description: An adverse event is considered "serious" if, in the view of either the investigator or sponsor, it results in any of the following outcomes:
  * Results in death,
  * Is life threatening,
  * Results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions,
  * Results in congenital anomaly, or birth defect,
  * Requires inpatient hospitalization or leads to prolongation of hospitalization
  * Other medically important events.
  Relationship to study drug was assessed by the investigator.
Time Frame: Up to 24 hours after study drug administration for each stress MPI (Day 1 and Day 2-15)
Population: Safety Analysis Set.
Measure: Number; unit: participants
Arm/Group | Regadenoson After Peak Exercise: MPI 1 | Regadenoson After Peak Exercise: MPI 2 | Regadenoson Alone: MPI 1 | Regadenoson Alone: MPI 2
Number analyzed (Participants) | 575 | 544 | 567 | 548
participants
  Any adverse event | 302 | 317 | 329 | 323
  Drug-related adverse event | 291 | 298 | 319 | 308
  Deaths | 0 | 0 | 0 | 0
  Serious adverse events | 5 | 2 | 1 | 1
  Drug-related serious adverse events | 2 | 0 | 0 | 0
  Adverse events leading to discontinuation | 13 | 0 | 5 | 1
  Drug-related AEs leading to discontinuation | 9 | 0 | 5 | 0

ADVERSE EVENTS:
Time Frame: From the time of administration of regadenoson to within 24 hours of administration of regadenoson for each stress MPI.
Arm/Group | Regadenoson After Peak Exercise: MPI 1 | Regadenoson After Peak Exercise: MPI 2 | Regadenoson Alone: MPI 1 | Regadenoson Alone: MPI 2
Serious Adverse Events (participants affected / at risk) | 5/575 | 2/544 | 1/567 | 1/548
Other Adverse Events (participants affected / at risk) | 277/575 | 274/544 | 307/567 | 290/548
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regadenoson After Peak Exercise: MPI 1 (N=575) | Regadenoson After Peak Exercise: MPI 2 (N=544) | Regadenoson Alone: MPI 1 (N=567) | Regadenoson Alone: MPI 2 (N=548)
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anticoagulation drug level below therapeutic (Investigations) | 0 | 0 | 0 | 1
Hepatic enzyme abnormal (Investigations) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Regadenoson After Peak Exercise: MPI 1 (N=575) | Regadenoson After Peak Exercise: MPI 2 (N=544) | Regadenoson Alone: MPI 1 (N=567) | Regadenoson Alone: MPI 2 (N=548)
Abdominal pain upper (Gastrointestinal disorders) | 31 | 35 | 35 | 34
Nausea (Gastrointestinal disorders) | 43 | 44 | 45 | 41
Chest discomfort (General disorders) | 37 | 33 | 54 | 43
Dizziness (Nervous system disorders) | 106 | 75 | 89 | 81
Headache (Nervous system disorders) | 85 | 108 | 137 | 118
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 141 | 125 | 161 | 152
Flushing (Vascular disorders) | 47 | 78 | 79 | 69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data or 18 months after data-lock, whichever is first. Sponsor must receive a site's manuscript at least 45 days prior to publication for review and comment. Sponsor may delay the publication for up to 60 days to seek patent protection.